CLINICAL TRIAL: NCT00281879
Title: Transplantation of Unrelated Donor Hematopoietic Stem Cells for the Treatment of Hematological Malignancies
Brief Title: Donor Stem Cell Transplant or Donor White Blood Cell Infusions in Treating Patients With Hematologic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard Maziarz, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000452794; P30CA016058 (NIH); OHSU-TPI-9695-L; OHSU-540
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Unusual Cancers of Childhood
Keywords: adult acute lymphoblastic leukemia in remission; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; L3 adult acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; L3 childhood acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); childhood acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; secondary acute myeloid leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia; chronic myelomonocytic leukemia; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL negative; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage III childhood Hodgkin lymphoma; stage III childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; unusual cancers of childhood; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Recurrence; Congenital Abnormalities; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Juvenile; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell | interventions — Antilymphocyte Serum; Filgrastim; Granulocyte Colony-Stimulating Factor; Busulfan; Carmustine; Cyclophosphamide; Cyclosporine; Cytarabine; Etoposide; fludarabine phosphate; Melphalan; Methotrexate; Methylprednisolone; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI) (Active Comparator)
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cyclosporine; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy
- Busulfan and Cyclophosphamide (Cytoxan) (Active Comparator)
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation
- BEAM Regimen (Active Comparator): On the day of your admission, you will start to take a drug called allopurinol which helps to protect your kidneys as your body works to discharge cells killed off by your chemotherapy and TBI. Chemotherapy will begin on Day -6 with carmustine (BCNU), followed by etoposide (VP-16), cytosine arabinoside (ARA-C), and melphalan. This conditioning regimen is known as the BEAM regimen. The dose of this therapy is high enough to kill cancer cells but will also kill all of your normal blood forming cells. Subjects undergoing the BEAM regimen will not have total body irradiation (TBI).
  Interventions: Biological: filgrastim; Drug: carmustine; Drug: cyclosporine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation
- Low-Dose Fludarabine and TBI(for second stem cell donation) (Active Comparator): A conditioning regimen of low-dose fludarabine and TBI is used in the event that a second donation of hematopoietic stem cells is necessary. Chemotherapy with Fludarabine will begin 4 days prior to your transplant. This drug will be given through the catheter in your chest daily for 3 days. TBI (radiation) will be given to you on the day of your transplant. After your TBI, your donor's stem cells / bone marrow will be given to you through your catheter. The drugs cyclosporine and mycophenolate mofetil (MMF) will be given orally to help you accept your donor's cells.
  Interventions: Biological: filgrastim; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy
- Busulfan, Cyclophosphamide, and Fludarabine (Pediatric only) (Active Comparator): On the day of your admission you will start to take a drug called Dilantin which is used to help prevent seizures while you receive your chemotherapy drugs. You will also start to take a drug called allopurinol which helps to protect your kidneys as your body works to discharge cells killed off by your chemotherapy and TBI. On the next day, you will then begin your conditioning therapy with a drug called busulfan. This medicine will be given to you by an infusion into your bloodstream through a small tube in the vein of your arm four times per day for four days. After the busulfan treatment, you will receive 4 doses each of two drugs, cyclophosphamide (also known as Cytoxan) and fludarabine, over 2 hours into your vein.
  Interventions: Biological: filgrastim; Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation
- ATG For Cord Blood Transplants (Active Comparator): If you are undergoing a pre-transplant conditioning regimen prior to undergoing a cord blood transplant, you will receive a drug called ATG to improve your chances of engraftment and decrease your risk of graft versus host disease. You may receive ATG 3 times during your transplant regimen on days -3 through days -1 in addition to your pre-transplant conditioning therapy. Methylprednisolone will also be given during each dose of ATG to help reduce any reactions during infusion.
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: cyclosporine; Drug: methotrexate; Drug: methylprednisolone; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation; Procedure: umbilical cord blood transplantation
- DLI (Donor Leukocyte Infusion) (Active Comparator): Donor Leukocyte Infusions: You will receive DLI from your original transplant donor. This will be given through a vein , usually in your arm. It will be similar to getting a platelet or blood transfusion. You may require more than one DLI. The decision to give you another infusion will be determined by your condition, relapse status, GVHD and how much DLI you were given before. You may need chemotherapy and/or radiation to improve your disease status prior to additional DLI's.
  Interventions: Biological: filgrastim; Drug: cyclosporine; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation
- Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric only) (Active Comparator): On the day after your admission, you will start receiving radiation therapy (TBI). Radiation will be given to you 2 times a day for 3 days. On the next day, you will then begin your chemotherapy with a drug called etoposide. This medicine will be given to you by an infusion into your bloodstream through a small tube in the vein of your arm for one day. After the etoposide treatment, on the next day you will receive cyclophosphamide (also known as Cytoxan) for 2 days. When you are given cyclophosphamide, you will also be given a medication called MESNA to help protect your bladder from damage. After you have completed the cyclophosphamide you will rest one day without any anti-cancer therapy. This allows your body time to remove and inactivate the chemotherapy. After a day of rest, you will be given your donor's cells.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cyclosporine; Drug: etoposide; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: anti-thymocyte globulin — Intravenous, 1.5 mg/kg of body weight daily for 7 to 14 days The first dose should be administered over a minimum of 6 hours and over at least 4 hours on subsequent doses through a high-flow vein.
  Other Names: ATG
  Arms: ATG For Cord Blood Transplants
Biological: filgrastim — Will be given IV at 5 µg/kg/day. The first injection will be administered on day +7, i.e. 7 days after the hematopoietic stem cells are infused.
  Will be administered until the ANC is 1500 / µl for 2 days. Dose and schedule of G-CSF administration is left to each center's discretion.
  Other Names: G-CSF
Drug: busulfan — Patients who take the drug PO, busulfan will be administered at 1 mg/kg/ dose given by mouth every 6 hours for 16 consecutive doses. Pediatric patients who receive busulfan IV continuous infusion will receive a dose of 3.0 mg/kg/IBW if under the age of 2.Pediatric patients over the age of 2 will receive busulfan at a dose of 0.8 mg/kg/dose.
  Arms: Busulfan and Cyclophosphamide (Cytoxan); Busulfan, Cyclophosphamide, and Fludarabine (Pediatric only)
Drug: carmustine — 300mg/m2 IV dissolved in 500 cc NS infused over 2 hours into right atrial catheter on day -6.
  Arms: BEAM Regimen
Drug: cyclophosphamide — For transplantation, the drug is diluted in 250 to 500 cc of NS or D5W and administered IV over 2 hours.
  Arms: Busulfan and Cyclophosphamide (Cytoxan); Busulfan, Cyclophosphamide, and Fludarabine (Pediatric only); Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI); Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric only)
Drug: cyclosporine — Initial doses will be administered IV at a starting dose of 1.5 mg/kg BID. The infusion will vary from 2-24hr depending on the incidence of side-effects.
Drug: cytarabine — 400 mg/m2 dissolved in 200cc D5W and infused over 30 minutes into right atrial catheter on days -5, -4, -3, -2.
  Arms: BEAM Regimen
Drug: etoposide — Etoposide administration 200 mg /m2 dissolved in 1 liter NS and infused over 2 hours into right atrial catheter. Infusion to begin after cytarabine administration on days -5, -4, -3, -2.
  Etoposide administration 50 mg/kg IV over 24 hours, divided into 3 doses. Dilute in normal saline at a concentration of 0.4 mg/ml (Observe for precipitation). Administered IV with continuous infusion over 24 hours. Diuretics may be given for fluid overload.
  Arms: BEAM Regimen; Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric only)
Drug: fludarabine phosphate — Fludarabine administered at 30 mg/m2 IVPB infused over 30 minutes into right atrial catheter on days -4, -3, -2.
  Fludarabine administered at 40 mg/m2 IVPB infused over 30 into the right atrial catheter on days -5, -4, -3, and -2.
  Arms: Busulfan, Cyclophosphamide, and Fludarabine (Pediatric only); Low-Dose Fludarabine and TBI(for second stem cell donation)
Drug: melphalan — 140 mg /m2 in concentration of 0.45 mg/ml of NS infused over 30 minutes into right atrial catheter on day -1.
  Arms: BEAM Regimen
Drug: methotrexate — Administered on days +1, +3, and +7.
Drug: methylprednisolone — Methyl-prednisolone is administered IV as a rapid infusion.
  Arms: ATG For Cord Blood Transplants
Drug: mycophenolate mofetil — Mycophenolate may be used as a substitute for Methotrexate
Drug: tacrolimus — A drug used to decrease the risk of graft versus host disease (GvHD).
  Other Names: FK-506
Procedure: peripheral blood stem cell transplantation — The stem cells will be given to you by intravenous injection (through your vein) using a catheter that was placed prior to beginning chemotherapy. The stem cell infusion takes 1-6 hours.
Procedure: umbilical cord blood transplantation — The patient will receive ATG to improve the changes of engraftment and decrease their risk of graft versus host disease. The patient may receive ATG 3 times during their transplant regimen on days -3 through days -1
  Arms: ATG For Cord Blood Transplants
Radiation: radiation therapy — Radiation will be given to you 2 times a day for 3 or 4 days.
  Arms: Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI); Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric only); Low-Dose Fludarabine and TBI(for second stem cell donation)

SUMMARY:
RATIONALE: A peripheral stem cell transplant or an umbilical cord blood transplant from a donor may be able to replace blood-forming cells that were destroyed by chemotherapy or radiation therapy. Giving an infusion of the donor's white blood cells (donor lymphocyte infusion) after the transplant may help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells can make an immune response against the body's normal cells. Methotrexate, cyclosporine, tacrolimus, or methylprednisolone may stop this from happening.

PURPOSE: This clinical trial is studying how well a donor stem cell transplant or donor white blood cell infusions work in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effectiveness of unrelated donor allogeneic hematopoietic stem cells for transplantation after conditioning for the treatment of patients with high-risk hematologic malignancies.
* Compare survival, disease-free survival (DFS), response rate, and toxicity rates in these patients with historical controls.
* Compare the rate and severity of acute and chronic GVHD after allogeneic hematopoietic stem cell transplantation in patients with hematopoietic malignancies with historical controls transplanted with stem cells from related sibling donors
* Assess engraftment, long-term hematopoietic recovery, relapse rate, and disease-free survival when allogeneic hematopoietic stem cells are used as a source of stem cells for transplantation in patients with high-risk hematological malignancies.
* Assess engraftment, long-term hematopoietic recovery, and overall survival when allogeneic hematopoietic stem cells are used as a source of stem cells for transplantation in patients who have graft failure or graft rejection.
* Compare engraftment, long-term hematopoietic recovery, rate of GVHD, rate of relapse, toxicity rates, overall disease-free survival and overall survival when donor leukocyte infusions (DLI) are given for patients who have disease recurrence, progression, or low donor chimerisms after unrelated stem cell transplantation or before DLI with historical controls of other donor leukocyte infusions.

Secondary

* Determine the quality of life of patients undergoing hematopoietic stem cell transplantation or donor leukocyte infusions from unrelated HLA genotypically-identical donors.

OUTLINE: Patients are assigned to 1 of 8 treatment groups.

* Group 1*: Patients undergo total body irradiation (TBI) twice a day on days -7 to -4. Patients then receive cyclophosphamide IV over 1 hour on days -3 and -2. On day 0 patients undergo stem cell transplantation (SCT). Beginning on day 7, patients receive filgrastim (G-CSF) IV once daily until blood counts recover.
* Group 2 (patients who have previously experienced dose-limiting radiotherapy): Patients receive oral busulfan 4 times daily on days -7 to -4 and cyclophosphamide IV over 1 hour on days -3 and -2. On day 0 patients undergo SCT. Beginning on day 7, patients receive G-CSF IV once daily until blood counts recover.
* Group 3 (pediatric patients only): Patients receive busulfan IV 4 times daily on days -9 to -6 and cyclophosphamide IV over 1 hour and fludarabine IV over 30 minutes on days -5 to -2. On day 0 patients undergo SCT. Beginning on day 7, patients may receive G-CSF IV once daily until blood counts recover.
* Group 4 (second SCT for patients who have experienced graft rejection or failure)*: Patients receive low-dose fludarabine IV over 30 minutes on days -4 to -2. Patients then undergo low-dose TBI once followed by SCT on day 0. Beginning on day 7, patients may receive G-CSF IV once daily until blood counts recover.
* Group 5 (patients who developed grade 3 cystitis after prior cyclophosphamide-containing therapy): Patients receive carmustine IV over 2 hours on day -6, etoposide IV over 2 hours and cytarabine IV over 30 minutes on days -5 to -2, and melphalan IV over 30 minutes on day -1 (BEAM). On day 0, patients undergo SCT. Beginning on day 7, patients receive G-CSF IV once daily until blood counts recover.
* Group 6 (cord blood transplantation): Patients receive anti-thymocyte globulin IV once daily and methylprednisolone IV twice daily on days -3 to -1. On day 0, patients undergo an umbilical cord blood SCT.
* Group 7 (patients with relapsing or progressive disease after prior transplants or low donor chimerisms)*: Patients must not have existing graft-versus-host disease (GVHD). Patients receive donor lymphocyte infusions with conditioning chemotherapy and/or radiotherapy at the discretion of the investigator.
* Group 8 (pediatric patients only)*: Patients undergo TBI twice a day on days -7 to -5. Patients also receive etoposide IV over 24 hours on day -4 and cyclophosphamide IV over 1 hour on days -3 and -2. On day 0, patients undergo SCT. Beginning on day 7, patients may receive G-CSF IV once daily until blood counts recover.

NOTE: *Patients who have received > 3000 cGy to the central nervous system or > 2000 cGy to the lung or liver may not receive any regimen containing total body irradiation (TBI)

All patients receive GVHD prophylaxis comprising methotrexate IV on days 1, 3, 6, and 11; cyclosporine and/or tacrolimus on days -2 to 100; and/or methylprednisolone IV on days 7 to 100.

Patients with an unrelated donor who experience a relapse prior to transplantation, may proceed directly to transplantation. However, if immediate transplantation from the unrelated donor is not possible, the patient must be re-induced into a complete hematological remission. Patients who experience graft failure or graft rejection after allogeneic transplantation are eligible for a second stem cell infusion from the original donor.

Quality of life is assessed at baseline and at 7 days, 3 months, and 1 year after transplantation.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following*:

  * Acute lymphoblastic leukemia in any disease phase

    * Patients with any of the following high-risk features are encouraged to enroll:

      * Philadelphia chromosome positive disease
      * L3 morphology, especially in the presence of t(8;14), t(8;22), or t(2;8)
      * Patients not in remission at day 28 of first induction
      * High LDH (i.e., ≥ 300 IU/mL at presentation)
      * Pre-B-cell, mixed lineage, or Burkitt's markers
      * Relapsed in the marrow while receiving continuous chemotherapy
      * Within 6 months after stopping chemotherapy
      * Relapse in one organ or extramedullary relapses in more than one organ while still receiving chemotherapy
  * Hodgkin's or non-Hodgkin's lymphoma beyond first complete remission (CR) or in first CR with features of high-risk disease, including, but not limited to:

    * Lymphoma not in CR after 3 courses of primary therapy
    * Patients with bulky disease at presentation, especially bulky mediastinal disease
    * Patients with LDH ≥ 300 IU/mL at presentation
    * Patients with extranodal disease
    * Patients with first remission within less than 1 year
    * Stage IV disease at presentation, especially with marrow involvement
    * Patients with high-intermediate or high International Index Scores
  * Acute myeloid leukemia (AML) meeting the following criteria:

    * Beyond first remission or high-risk disease in first CR
    * Required multiple courses of induction therapy to achieve a remission
    * Had residual leukemia on day 14-28 bone marrow examination after initial induction
    * Patients with any cytogenetic abnormality except inv 16 or t(8;21)
  * Chronic myelogenous leukemia in the chronic or early accelerated phase of the disease

    * Patients with blast crisis that can be induced back into chronic phase may be transplanted in second chronic phase
  * Myelodysplastic syndromes (MDS) meeting the following requirements:

    * Transfusion-dependent refractory anemia (RA), RA with excess blasts (RAEB), RAEB in transformation, or chronic myelomonocytic leukemia (CMML)
    * Patients with MDS that present with or evolve to AML must be re-induced back to remission prior to initiating a search for an unrelated donor NOTE: *Patients with other hematologic malignancies not listed above, including diseases such as chronic lymphocytic leukemia (CLL), multiple myeloma, or rare pediatric malignancies, or patients who are felt to be at high-risk for relapse but who do not have features listed, may be allowed at the discretion of the investigator.
* Must have failed prior stem cell transplantation
* Must have a suitable unrelated allogeneic hematopoietic stem cell donor

  * A 5/6 match degree is acceptable for unrelated bone marrow donors
  * A 4/6 match degree is acceptable for unrelated cord blood units

PATIENT CHARACTERISTICS:

* SWOG performance status (PS) 0-2 OR
* Karnofsky PS 50-100% OR
* Lansky PS 50-100%
* Creatinine clearance ≥ 45 mL/min
* Creatinine ≤ 2.5 mg/dL
* Bilirubin ≤ 2 mg/dL (abnormally high liver function tests allowed if the only source for the elevation is due to lymphoma of the liver)
* AST or ALT ≤ 2 times normal (abnormally high liver function tests allowed if the only source for the elevation is due to lymphoma of the liver)
* No patients at high risk of veno-occlusive disease
* Not pregnant or nursing
* Negative serum pregnancy test
* Fertile patients must use an effective contraceptive method
* DLCO ≥ 50% of predicted
* FEV_1/FVC ≥ 65% of predicted
* No current congestive heart failure (CHF) and/or LVEF ≥ 45%
* No myocardial infarction within the past 6 months
* No unstable angina within the past 6 months
* HIV negative
* Life expectancy must not be limited by disease other than malignancy
* No allergy to any chemotherapeutic agent included in the regimen

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Maziarz, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI): On admission day, you will start to take a drug called allopurinol which helps to protect your kidneys as your body works to discharge cells killed off by your chemotherapy and TBI. Allopurinol tablets will be given to you by mouth up to three times a day for 7 days. You will begin radiation therapy to your entire body at the start of your transplant treatment. This procedure is called TBI (total body irradiation). Radiation will be given to you 2 times a day for 3 or 4 days. After the radiation treatment, you will receive two doses of cyclophosphamide by vein (through a small plastic tube leading into the bloodstream). Each dose takes about 2 hours to administer. When you are given cyclophosphamide, you will also be given a medication called MESNA to help protect your bladder from damage. After you have completed the cyclophosphamide you will rest one day without any anti-cancer therapy.
- Busulfan and Cyclophosphamide (Cytoxan): On admission day, you will start to take a drug called Dilantin, which is used to help prevent seizures while you receive your chemotherapy drugs. You will also start to take a drug called allopurinol,which helps to protect your kidneys as your body works to discharge cells killed off by your chemotherapy and TBI. Allopurinol tablets will be given to you by mouth up to three times a day for 7 days. You will begin the therapy with a drug called busulfan. This medicine is take by mouth four times per day for four days. After the oral busulfan treatment, you will receive two doses of cyclophosphamide over 2 hours by vein (through a small tube leading into the bloodstream). When you are given cyclophosphamide, you will also be given a medication called MESNA to help protect your bladder from damage. Subjects undergoing the Busulfan and Cyclophosphamide regimen will not have total body irradiation (TBI).
Period: Overall Study
Arm/Group | Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI) | Busulfan and Cyclophosphamide (Cytoxan) | BEAM Regimen | Low-Dose Fludarabine and TBI(for Second Stem Cell Donation) | Busulfan, Cyclophosphamide, and Fludarabine (Pediatric Only) | ATG For Cord Blood Transplants | DLI (Donor Leukocyte Infusion) | Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric Only)
Started | 128 | 36 | 20 | 0 | 6 | 9 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 128 | 36 | 20 | 0 | 6 | 9 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI) | Busulfan and Cyclophosphamide (Cytoxan) | BEAM Regimen | Low-Dose Fludarabine and TBI(for Second Stem Cell Donation) | Busulfan, Cyclophosphamide, and Fludarabine (Pediatric Only) | ATG For Cord Blood Transplants | DLI (Donor Leukocyte Infusion) | Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric Only) | Total
Number analyzed (Participants) | 128 | 36 | 20 | 0 | 6 | 9 | 0 | 1 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 1 | 0 |  | 6 | 7 |  | 1 | 42
  Between 18 and 65 years | 101 | 35 | 20 |  | 0 | 0 |  | 0 | 156
  >=65 years | 0 | 0 | 0 |  | 0 | 2 |  | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.033 (14.923) | 48.33 (11.67) | 46.187 (12.87) |  | 12.22 (7.90) | 11.77 (10.725) |  | 5.42 (0) | 34.743 (16.818)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 13 | 3 |  | 4 | 5 |  | 1 | 82
  Male | 72 | 23 | 17 |  | 2 | 4 |  | 0 | 118
Region of Enrollment [Number; unit: participants]
  United States | 128 | 36 | 20 |  | 6 | 9 |  | 1 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Free Survival (DFS).
Description: Determine the effectiveness of unrelated donor allogeneic hematopoietic stem cells for transplantation after conditioning for the treatment of high-risk hematopoietic malignancies.
  Disease-free survival: The length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer.
Time Frame: Duration of the study; Up to 2 years
Arm/Group | Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI) | Busulfan and Cyclophosphamide (Cytoxan) | BEAM Regimen | Low-Dose Fludarabine and TBI(for Second Stem Cell Donation) | Busulfan, Cyclophosphamide, and Fludarabine (Pediatric Only) | ATG For Cord Blood Transplants | DLI (Donor Leukocyte Infusion) | Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric Only)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI) | Busulfan and Cyclophosphamide (Cytoxan) | BEAM Regimen | Low-Dose Fludarabine and TBI(for Second Stem Cell Donation) | Busulfan, Cyclophosphamide, and Fludarabine (Pediatric Only) | ATG For Cord Blood Transplants | DLI (Donor Leukocyte Infusion) | Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric Only)
Serious Adverse Events (participants affected / at risk) | 101/128 | 25/36 | 17/20 | 0/0 | 5/6 | 6/9 | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 19/128 | 0/36 | 2/20 | 0/0 | 0/6 | 0/9 | 0/0 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI) (N=128) | Busulfan and Cyclophosphamide (Cytoxan) (N=36) | BEAM Regimen (N=20) | Low-Dose Fludarabine and TBI(for Second Stem Cell Donation) (N=0) | Busulfan, Cyclophosphamide, and Fludarabine (Pediatric Only) (N=6) | ATG For Cord Blood Transplants (N=9) | DLI (Donor Leukocyte Infusion) (N=0) | Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric Only) (N=1)
Staph Sepsis (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Altered mental status (Psychiatric disorders) | 1 | 1 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Death (General disorders) | 101 | 25 | 17 | 0 (0) | 5 | 6 | 0 (0) | 1 (1)
Fever (Immune system disorders) | 0 | 0 | 1 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Graft versus host disease (GVHD) (Gastrointestinal disorders) | 17 | 13 | 3 | 0 (0) | 1 | 0 | 0 (0) | 0 (0)
Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0 (0) | 1 | 0 | 0 (0) | 1
Cardiac Problems (Cardiac disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Diarrhea (General disorders) | 4 | 2 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Orthostatic Hypertension (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
acute renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 0 (0) | 0 | 0 | 0 (0) | 1
Intraparenchymal Hemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 (0) | 1 | 0 | 0 (0) | 0 (0)
Rigors (Immune system disorders) | 3 | 2 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Pneutropenic Fever (Immune system disorders) | 3 | 2 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Kidney Stones (Renal and urinary disorders) | 0 | 3 | 2 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Encephalopathy (Infections and infestations) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Viral encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Pulmonary aspergillus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Anorexia (Psychiatric disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Dehydration (General disorders) | 3 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 15 | 3 | 2 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Bacterial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Seizures (General disorders) | 2 | 1 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Cytomegalovirus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Positive blood cultures (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 | 1 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Liver failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 (0) | 0 | 0 | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 11 | 2 | 2 | 0 (0) | 0 | 1 | 0 (0) | 0 (0)
Steroid-induced psychoses (Psychiatric disorders) | 1 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide (Cytoxan) and Total Body Irradiation (TBI) (N=128) | Busulfan and Cyclophosphamide (Cytoxan) (N=36) | BEAM Regimen (N=20) | Low-Dose Fludarabine and TBI(for Second Stem Cell Donation) (N=0) | Busulfan, Cyclophosphamide, and Fludarabine (Pediatric Only) (N=6) | ATG For Cord Blood Transplants (N=9) | DLI (Donor Leukocyte Infusion) (N=0) | Cyclophosphamide, Etoposide (VP16) and TBI (Pediatric Only) (N=1)
Headache (General disorders) | 8 | 0 | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (General disorders) | 11 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No